CLINICAL TRIAL: NCT04633096
Title: The Efficacy of Automated Feedback After Internet-based Depression Screening: the German, Three-armed, Randomised Controlled Trial DISCOVER
Brief Title: The Efficacy of Automated Feedback After Internet-based Depression Screening
Acronym: DISCOVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Dr. Sebastian Kohlmann, Senior Researcher, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Screening
Other Study IDs: PV7039
Record Dates: First submitted 2020-11-06; First posted 2020-11-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Depression; Major Depressive Disorder
Keywords: Depression; Screening; Tailored feedback; Internet-based intervention; Early Detection
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tailored feedback (Experimental): Using a randomized-controlled study design one third of the participants will receive individually tailored feedback after depression screening. The feedback for the participant contains the screening result, information about depression in general, guideline based treatment recommendations for patients and contact-information for treatment. The information is tailored to the participant's individual symptom profile, illness perceptions and preferences.
  Interventions: Behavioral: tailored feedback of depression screening results
- standardized feedback (Experimental): Using a randomized-controlled study design one third of the participants will receive a standard feedback after depression screening. The feedback for the participant contains the screening result, information about depression in general, guideline based treatment recommendations for patients and contact-information for treatment.
  Interventions: Behavioral: standardized feedback of depression screening results
- no feedback (No Intervention): Using a randomized-controlled study design one third of the participants will not receive any feedback.

INTERVENTIONS:
Behavioral: tailored feedback of depression screening results — The feedback for the participant contains the screening result, information about depression in general, guideline based treatment recommendations for patients and contact-information for treatment. The information is tailored to the participant's individual symptom profile, illness perceptions and preferences.
  Arms: tailored feedback
Behavioral: standardized feedback of depression screening results — The feedback for the participant contains the screening result, information about depression in general, guideline based treatment recommendations for patients and contact-information for treatment.
  Arms: standardized feedback

SUMMARY:
The DISCOVER randomized controlled trial is designed to evaluate the effect of automated feedback after internet-based depression screening in individuals with undetected depression. A total of 1076 individuals reporting elevated levels of depression (PHQ-9 score ≥ 10 points) will be randomized into three groups to either receive a) no feedback (control group), b) standardised or c) tailored feedback on their depression screening results.The primary hypothesis is that feedback reduces depression severity six months after screening compared to no feedback. The secondary hypothesis is that tailored feedback is more efficacious as compared to standard feedback.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a highly prevalent condition associated with substantial disease burden and economic costs. Still, it often remains undetected and untreated, which in turn increases the likelihood of a chronic course, treatment resistance and rising healthcare costs. One solution to address early detection and disease burden could be widely accessible depression screening. Our previous trial in cardiac patients provides first evidence that depression screening combined with written individual-targeted feedback on the screening results improves depression severity and encourages greater patient participation and engagement in mental health. To amplify these effects in a broader setting, the internet-based DISCOVER randomized controlled trial (RCT) now aims at addressing affected but yet undetected individuals on the internet. In order to evaluate the effect of feedback in this setting, a total of 1076 individuals reporting elevated levels of depression (PHQ-9 score ≥ 10) will be randomized into three groups. They either receive a) no feedback (control group), b) standardised or c) tailored feedback on their depression screening results. The primary hypothesis is that feedback reduces depression severity six months after screening compared to no feedback. The secondary hypothesis is that tailored feedback is more efficacious as compared to standard feedback. Futher outcomes are guideline-based depression care, depression-related help-seeking behaviour, a health economic evaluation, clinical outcomes (somatic symptom severity and anxiety), health-related quality of life, illness beliefs, intervention acceptance, depression diagnosis and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* (Gender: male, female, diverse)
* Age ≥ 18 years; no maximum age
* Sufficient German language skills
* Informed consent
* Patient Health Questionnaire-9 > 9 points
* Contact details
* Internet access
* Sufficient computer/internet literacy

Exclusion Criteria:

* Diagnosis of a depressive disorder within the past 12 months
* Depression treatment (current or within the past 12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1178 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Depression severity (Questionnaire: Patient Health Questionnaire-9) | Six months after screening
  Level of depression severity assessed six months after screening with the Patient Health Questionnaire-9. Score range is 0 to 27 points. Higher scores mean more severe depression.

SECONDARY OUTCOMES:
Depression severity (Questionnaire: Patient Health Questionnaire-9) | One month after screening
  Level of depression severity assessed one month after screening with the Patient Health Questionnaire-9. Score range is 0 to 27 points. Higher scores mean more severe depression.
Guideline-based depression care | Six months after screening
  Proportion of individuals treated according to German Guideline based recommendations (e.g. depression diagnosis by a health professional, psychotherapy)
Depression-related help-seeking behaviour | Six months after screening
  proportion of individuals seeking formal and informal help, including information seeking, self-help, online help, professional help.
Health economic Evaluation (Questionnaire: Client Sociodemographic and Service Receipt Inventory) | Six months after screening
  Health care use assessed six months after screening with the Client Sociodemographic and Service Receipt Inventory. The Client Sociodemographic and Service Receipt Inventory assesses health care use by assessing the use of healthcare services (e.g. hospital stays, health professional contacts), medication (e.g. type of drug) and work loss days (e.g. hospital days)
Health-related quality of life (Questionnaire: EuroQol-5D) | Six months after screening
  Health-related quality of life assessed six months after screening with the EuroQol-5D. The EuroQol-5D (EQ5D) consists of five items with a 4 point Likert scale reflecting five different dimensions of quality of life. Higher scores reflect better quality of life.
Anxiety (Questionnaire: Generalized Anxiety Disorder-7) | Six months after screening
  Level of anxiety assessed six months after screening with the Generalized Anxiety Disorder-7. Score range is 0 to 21 points. Higher scores mean more anxiety.
Somatic symptom severity (Questionnaire: Somatic Symptom Scale-8) | Six months after screening
  Level of somatic symptom severity assessed six months after screening with the Somatic Symptom Scale.8. Score range is 0 to 32 points. Higher scores mean more somatic symptom burden.
Intervention acceptance (Questionnaire: Usefulness scale for patient information material) | One month after screening
  Usefulness and satisfaction with the feedback intervention material will be assessed one month after screening with the Usefulness Scale for patient information material. Score range is 0 to 100 points. Higher scores mean better usefulness. Items are added to assess PHQ-9-based depression screening.
Adverse events | Six months after screening
  Proportion of individuals reporting the occurence of any negative event that is attributed to the trial assessed by one open question six months after screening

OTHER OUTCOMES:
Illness beliefs (Questionnaire: Brief-Illness Perception Questionnaire) | One and six months after screening
  Depression-related illness beliefs assessed one and six months after screening with the Brief-Illness Perception Questionnaire. The Brief-Illness Perception Questionnaire includes 8 subscales (consequences, timeline, personal control, treatment control, illness comprehensibility, illness concern, illness-related emotions, causal attribution). Depending on each scale higher scores can represent functional or dysfunctional illness representations.
Depression Diagnosis (Structured Clinical Interview for DSM-5 Disorders; depression-related module) | Two days and six months after screening
  Proportion of individuals with a depression diagnosis as assessed with the Structured Clinical Interview for DSM-5 Disorders (depression-related module)
Critical life events | Six months after screening
  Positive and negative critical life events, assessed by open questions six months after screening
Website use | At baseline
  Number of clicks per page
Intervention adherence | Six months after screening
  Extent to which participants have read the feedback (in percentage), as reported by participants six months after screening

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Kohlmann, PhD, Principal Investigator — University Medical Center Hamburg-Eppendorf, Department of Psychosomatic Medicine and Psychotherapy
Locations (1):
- University Medical Center Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the ethics approval of the Ethics Committee of the Hamburg Medical Association on 29 July 2019, (approval number PV7039) and the German Research Foundation guidelines for the handling of research data, deidentified data will be made available on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available six months after publication of the main findings. Data will be available for ten years after publication of the main findings.
Access Criteria: Data can be requested by the principal investigators. Data use and request are subject to the publication policy of the DISCOVER RCT.

REFERENCES:
- [Background] Sikorski F, Konig HH, Wegscheider K, Zapf A, Lowe B, Kohlmann S. The efficacy of automated feedback after internet-based depression screening: Study protocol of the German, three-armed, randomised controlled trial DISCOVER. Internet Interv. 2021 Jul 21;25:100435. doi: 10.1016/j.invent.2021.100435. eCollection 2021 Sep. PMID 34401394
- [Derived] Sikorski F, Lowe B, Daubmann A, Kohlmann S. Potential Harms of Feedback After Web-Based Depression Screening: Secondary Analysis of Negative Effects in the Randomized Controlled DISCOVER Trial. J Med Internet Res. 2025 Apr 30;27:e59476. doi: 10.2196/59476. PMID 40305104
- [Derived] Kohlmann S, Sikorski F, Konig HH, Schutt M, Zapf A, Lowe B. The efficacy of automated feedback after internet-based depression screening (DISCOVER): an observer-masked, three-armed, randomised controlled trial in Germany. Lancet Digit Health. 2024 Jul;6(7):e446-e457. doi: 10.1016/S2589-7500(24)00070-0. PMID 38906611
- See also: Study protocoll — https://doi.org/10.1016/j.invent.2021.100435

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT04633096/SAP_000.pdf